CLINICAL TRIAL: NCT00571350
Title: Anterior Vaginal Wall Reconstruction: Anterior Colporrhaphy Reinforced With Tension Free Vaginal Tape Underneath Bladder Base
Brief Title: Anterior Vaginal Wall Reconstruction
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Hippocration General Hospital (Other)
Responsible Party: 2nd OBSTETRICS AND GYNECOLOGY UNIVERSITY CLINIC, HIPPOKRATIO UNIVERSITY HOSPITAL
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: ARISFC; HIPPOKRATIO HOSPITAL
Record Dates: First submitted 2007-12-10; First posted 2007-12-12 (Estimated); Last update posted 2007-12-12 (Estimated); Status verified 2007-12

CONDITIONS: Vaginal Prolapse
Keywords: Cystocele; tension free vaginal tapes; urinary incontinence
MeSH Terms: conditions — Uterine Prolapse; Cystocele; Urinary Incontinence

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- A (Active Comparator): women with vaginal prolapse who underwent TVT O
  Interventions: Procedure: tvt-o operation; Procedure: tvt o operation

INTERVENTIONS:
Procedure: tvt-o operation — transvaginal tention free obturator tape
  Other Names: Johnson & Johnson Ethicon Gyneacare, Somerville, NJ, USA
Procedure: tvt o operation — transobturator vaginal tape insertion
  Other Names: tention free vaginal tape

SUMMARY:
The purpose of this study is to assess the effectiveness of the polypropylene tape in preventing cystocele recurrence when placed underneath the bladder base as a concomitant measure to the anterior colporrhaphy procedure.

DETAILED DESCRIPTION:
Objective: The purpose of this study is to assess the effectiveness of the polypropylene tape in preventing cystocele recurrence when placed underneath the bladder base as a concomitant measure to the anterior colporrhaphy procedure.

Methods: Fifty Caucasian women 50 to 77 years old (mean age 66.6 years), 2 pre and 48 post menopausal with stage II-IV pelvic organ prolapse, enrolled into the study. Vaginal reconstructive surgery included an anterior colporrhaphy in all patients, posterior colpoperineorrhaphy in 28 patients and hysterectomy in 36 patients. They were randomly divided in a control group of 22 women and a study group of 28 women. As reinforcement to the anterior colporrhaphy procedure a polypropylene tape (TVT-O) was placed not under the midurethra, as originally described in case of stress incontinence, but underneath the bladder base and was fixed there with polyglactin sutures, in the study group. The postoperative follow up was carried out in frequent intervals of 4 months (total 48 months). The assessment of the anatomic result included evaluation of the operated sites and of the position of the tapes inserted on clinical grounds and after perineal sonography, which measured the distance of the bladder base to the inferior edge of the symphysis pubis.

Results: In all patients the postoperative correction of the anterior vaginal wall was sufficient; the mean distance of the bladder base to the inferior edge of the symphysis pubis was 1.5 cm (range 1.0-2.2 cm). Mean residual urine volume was 30 ml. There were postoperatively 2 cases of stress incontinence and two cases of urge incontinence one in each group. There was no case of tape erosion noted, no dyspareunia and no recurrent cystocele in the study group. Four cases of recurrent cystocele (20%) were reported in our control group.

Conclusion: The tension free vaginal tape, particularly TVT-O, placed underneath the bladder base, when performed concomitantly to the anterior colporrhaphy appears to be safe and effective. While the preliminary results of our study are encouraging, larger series of patients and longer follow up are required to verify the effectiveness of the aforementioned modification.

ELIGIBILITY:
Inclusion Criteria:

* Women 50-77 years old with stage II-IV organ prolapse

Ages: 50 Years to 77 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2005-01; Study Completion 2007-12 (Estimated)

PRIMARY OUTCOMES:
The purpose of this study is to assess the effectiveness of the polypropylene tape in preventing cystocele recurrence when placed underneath the bladder base as a concomitant measure to the anterior colporrhaphy procedure. | 2008

SECONDARY OUTCOMES:
GOOD QUALITY OF LIFE FOR PATIENTS | 2008

CONTACTS AND LOCATIONS:
Overall Officials: ANGELOS DANIILIDIS, MD, Principal Investigator — HIPPOKRATIO UNIVERSITY HOSPITAL; JOHN TZAFETTAS, PROFESSOR, Study Director — HIPPOKRATIO UNIVERSITY HOSPITAL; THEOHARIS TANTANASIS, ASS PROF, Principal Investigator — HIPPOKRATIO UNIVERSITY HOSPITAL
Locations (1):
- Medical School Aristotle University, Thessaloniki, Greece

REFERENCES:
- [Background] Sand PK, Koduri S, Lobel RW, Winkler HA, Tomezsko J, Culligan PJ, Goldberg R. Prospective randomized trial of polyglactin 910 mesh to prevent recurrence of cystoceles and rectoceles. Am J Obstet Gynecol. 2001 Jun;184(7):1357-62; discussion 1362-4. doi: 10.1067/mob.2001.115118. PMID 11408853